CLINICAL TRIAL: NCT05683782
Title: ''Erythropoietin Gel as an Adjunct to Split-Thickness Apically Positioned Flap in Augmentation of Attached Gingiva'' (A Randomized Controlled Clinical Study)
Brief Title: Erythropoietin Gel as an Adjunct to Split-Thickness Apically Positioned Flap in Augmentation of Attached Gingiva
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Fadl, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erythropoietin Gel
Record Dates: First submitted 2022-03-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Erythropoietin; Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test Group (Active Comparator): Split-thickness Apically Positioned Flap with topical Erythropoietin (Test group):
  A split thickness horizontal incision will be done at the mucogingival junction of the targeted area to be augmented with a scalpel with blade number 15C. Around the teeth, the gingiva stays intact coronal to the horizontal incision. The horizontal incision will extend mesio-distally in accordance with the area to be augmented.(Mandibular anterior or premolar teeth).
  A split-thickness flap is elevated, and the dissection is extended as far as necessary in the apical direction. The flap is secured to the periosteum with simple interrupted bio absorbable sutures.
  A Chitosan based Erythropoietin gel will be prepared. 1 mL of EPO-loaded with chitosan 5% and β-glycerophosphate disodium salt (GP) 20% gel will be used. The patient will be instructed to use the gel on the surgical site two times daily for 14 days.
  Interventions: Drug: Split thickness Apically positioned flap with Chitosan based Erythropoietin Gel application
- Control Group (Active Comparator): Split-thickness Apically Positioned Flap without Erythropoietin :
  Local anesthesia is administered by infiltration technique. The same surgical procedure is performed with the application of Chitosan gel without being loaded with erythropoietin.
  Interventions: Drug: Split thickness Apically positioned flap without Erythropoietin application

INTERVENTIONS:
Drug: Split thickness Apically positioned flap with Chitosan based Erythropoietin Gel application — Split thickness Apically positioned flap will be performed to increase width of attached gingiva .1 mL of EPO-loaded with chitosan 5% and β-glycerophosphate disodium salt (GP) 20% gel will be used by the patient two times daily for 14 days.
  Arms: Test Group
Drug: Split thickness Apically positioned flap without Erythropoietin application — Split thickness Apically positioned flap will be performed to increase width of attached gingiva.The patient will use a Chitosan gel without being loaded with erythropoietin two times daily for 14 days
  Arms: Control Group

SUMMARY:
This study will be carried out to evaluate the effect of topical application of erythropoietin gel as an adjunct to split-thickness apically positioned flap regarding Wound Healing and the Effect on post-surgical symptoms [ Patient Satisfaction] (1ry objective) and Clinical gain in width of attached gingiva. (2ry objective).

DETAILED DESCRIPTION:
The gingiva is divided into three parts anatomically: marginal, attached, and interdental. Attached gingiva, as defined by Orban, is the part of the gingiva that is firmly attached to the underlying tooth and bone and is stippled on the surface.

From the base of the gingival crevice to the mucogingival junction, lays the attached gingiva which is the firm resilient component of the gingiva. Through connective tissue, it is closely adhered to the underlying periosteal tissues of alveolar bone. To stabilize the marginal gingiva and resist external harm, an adequate zone of attached gingiva is required.

Lang proposed in 1972 that periodontal tissues require at least 2 mm of attached gingiva to maintain their health and survive the functional pressures of mastication and tooth cleaning. Gingival recession can be exacerbated by insufficient width or thickness of attached gingiva.

Many surgical procedures, such as apically positioned flaps, connective tissue grafts, and free gingival grafts, have been described to enhance the width of attached gingiva.

The apically positioned flap was one of the strategies that allowed surgeons to preserve and extend the width of attached gingiva. Two vertical incisions are made to release a complete full-thickness flap of gingiva and alveolar mucosa. The gingiva, alveolar mucosa, periosteum, and all structures within this flap are all shifted apically and sutured into place so that the flap's margin just covers the alveolar crests. With this surgical procedure, there was a risk of crestal bone resorption and additional attachment loss.

Carnio introduced a modified approach in 1999 to decrease the possibility of recession and attachment loss associated with the traditional apically positioned flap. The split-thickness flap used in this technique differs from the original in that the coronal aspect of the keratinized tissue is not separated from the tooth.

It is a useful method for increasing the width of attached gingiva by exposing the periosteum in the area where gingival augmentation is needed. Because there is no palatal donor tissue, this partial thickness flap elevation reduces the danger of recession and crestal bone loss, has low morbidity, and has a predictable tissue color match. The surgical site is completely encompassed by keratinized tissue, which acts as a source of keratinized tissue cells.

Secondary intention healing takes place by passing through four stages: Blood Clot formation, Inflammation, Granulation tissue formation and, Epithelialization. The blood clot formed contains large numbers of microorganisms that are phagocytized by polymorph nuclear leukocytes which migrates to the area in large numbers. Macrophages multiply, engulfing RBCs and dissolving PMNs. During healing, the source of granulation tissue is the retained periosteal connective tissue, the periodontal ligament, and the surrounding gingival tissues and lining mucosa. Epithelial cells start to migrate from the surrounding tissues. These cells move along a fibrin network. It can take up to 14 days for surface epithelialization to occur.

The split-thickness apically positioned flap has several advantages over other procedures, including low morbidity due to the lack of a second surgical site, less tissue handling, quicker operative time, good color match, good aesthetics, and no risk of postoperative recession. A key drawback of this procedure is that at least 0.5 mm of attached gingiva must be present clinically in order for the wound to be completely encompassed by keratinized tissue, which aids in the production of keratinized tissue in the surgical site.

Erythropoietin (EPO) is a glycoprotein hormone produced predominantly by the kidney that regulates the synthesis of red blood cells. The mature protein is made up of a 165-amino-acid polypeptide chain that is highly glycosylated at three N-linked and one O-linked glycosylation sites, resulting in a molecular mass of 30-34 kDa.

EPO is a pleiotropic factor with anti-apoptotic and cytoprotective properties in a variety of tissues. EPO receptors have been found on a variety of cells, including fibroblasts, macrophages, mast cells, and melanocytes. EPO boosts the production of vascular endothelial growth factor (VEGF) and speeds up the angiogenesis, granulation tissue creation, and collagen formation processes in the dermis.

In both acute and chronic tissue injury, erythropoietin has shown to have restorative effects. EPO promotes healing and function restoration by inhibiting pro-inflammatory cytokines such as TNF-α, IL-1 β, IL-6, IL-12, and IL-23 at the local level. The US Food and Drug Administration (FDA) approved recombinant human erythropoietin (EPO) for the treatment of anemia in patients with chronic renal disease and chemotherapy-associated anemia. It not only decreases the formation of reactive oxygen species and membrane lipid peroxidase, but also inhibits the synthesis of pro-inflammatory cytokines.

In 2017, Hosseinjani et al. investigated the effects of EPO mouthwash (50 IU/ml, 15 ml four times a day) on the healing of oral mucositis in a randomized controlled clinical trial. The mouthwash decreased the severity and duration of the oral mucositis lesions.

In 2018, Yaghobee showed that applying EPO to surgical palatal wounds had a healing effect. Because the oral mucosa's basal cells also express erythropoietin receptors, topical erythropoietin treatment was thought to be useful in treating oral lesions. 4,000 IU EPO was mixed with 1 mL of 3 percent hydroxyl ethyl cellulose to make EPO-containing gels.

Although mouthwash local therapy improved the healing of oral mucositis lesions, the anatomical features of the mouth and the washing effect of saliva in the oral cavity result in a short retention time for mouthwashes and other conventional liquid dosage forms, resulting in a short-lasting effect and low therapeutic efficacy of active medications.

For their unique characteristic of sol-gel transition in response to environmental stimuli such as temperature, pH, or ionic strength, environmentally responsive hydrogels have piqued interest in drug delivery and other biological sectors. As a result, these hydrogels can be easily supplied as a solution that swells and gels very quickly after administration. Due to the reduced frequency of medication administration, the so-formed gel will have the advantage of longer drug release in the surrounding medium, which will increase patient compliance.

A randomized controlled trial was conducted to determine the safety and efficacy of a topical EPO-containing gel as an additional therapy to standard-of-care (SOC) in the treatment of diabetic foot ulcers. Following daily treatment of DFUs with the EPO-containing gel, no side effects were observed. For the treatment of DFUs, topical EPO can be a safe and effective option.

The combination of erythropoietin gel on the split-thickness apically positioned flap in an attempt to benefit from its regenerative and healing capacity is a good point of research. To measure the gel's effect on tissue keratinization, attached gingival gain and controlling post-operative pain is our point of concern.

ELIGIBILITY:
Inclusion Criteria:

* Males and females within age range of 20-40 years.
* Patients free of systemic diseases according to Burket's oral health history questionnaire .
* Patients who can follow and maintain oral hygiene instructions.
* Patients having insufficient width of attached gingiva (<2mm) in labial aspect of lower anterior or premolar teeth and Miller Class I recession .
* Thick gingival phenotype.

Exclusion Criteria:

* Smokers.
* Pregnant and lactating females
* Unwillingness or inability to return for follow-up appointments
* High frenum attachment
* Crowding of test site teeth
* Vulnerable patients (those with mental or physical impairments).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 21 days
  Using toluidine blue epithelialization test to asses the wound healing. The surgical site will be stained with toluidine blue stain. The darkly stained bluish patches will be interpreted as wound sites that are still healing and have insufficient surface epithelialization. The darkly stained areas will be photographed and then uploaded to a picture editing software to determine their surface area using digital tracing.
Patient Satisfaction | 1 month
  By using a 10 cm horizontal visual analogue scale. The patients will be asked to rate the degree of pain Zero represents the least amount of pain and ten represents the most amount of pain.

SECONDARY OUTCOMES:
Width of Attached Gingiva | 1 month
  The width of attached gingiva is calculated 1 month after the surgery by subtracting the pocket depth from total width of gingiva till the mucogingival junction.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Amr, Assoc.Prof, Study Director — Ain Shams University; Hala k Abdelgaber, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Yaghobee S, Rouzmeh N, Taheri M, Aslroosta H, Mahmoodi S, Mohammadnejad Hardoroodi M, Soleimanzadeh Azar P, Khorsand A. Evaluation of topical erythropoietin application on the healing outcome of gingival graft recipient site; a randomized controlled clinical trial. BMC Oral Health. 2021 Nov 12;21(1):578. doi: 10.1186/s12903-021-01948-8. PMID 34772399
- [Background] Yaghobee S, Rouzmeh N, Aslroosta H, Mahmoodi S, Khorsand A, Kharrazifard MJ. Effect of Topical Erythropoietin (EPO) on palatal wound healing subsequent to Free Gingival Grafting (FGG). Braz Oral Res. 2018 Jun 11;32:e55. doi: 10.1590/1807-3107bor-2018.vol32.0055. PMID 29898030
- [Background] Rezazadeh M, Jafari N, Akbari V, Amirian M, Tabbakhian M, Minaiyan M, Rostami M. A mucoadhesive thermosensitive hydrogel containing erythropoietin as a potential treatment in oral mucositis: in vitro and in vivo studies. Drug Deliv Transl Res. 2018 Oct;8(5):1226-1237. doi: 10.1007/s13346-018-0566-9. PMID 30076521
- [Background] Hamed S, Belokopytov M, Ullmann Y, Safadi M, Stark Y, Shoufani A, Akita S, Liu PY, Teot L. Interim Results of the Remede d'Or Study: A Multicenter, Single-Blind, Randomized, Controlled Trial to Assess the Safety and Efficacy of an Innovative Topical Formulation of Erythropoietin for Treating Diabetic Foot Ulcers. Adv Wound Care (New Rochelle). 2019 Oct 1;8(10):514-521. doi: 10.1089/wound.2018.0808. Epub 2019 Aug 21. PMID 31832270
- [Background] Brines M, Cerami A. Erythropoietin-mediated tissue protection: reducing collateral damage from the primary injury response. J Intern Med. 2008 Nov;264(5):405-32. doi: 10.1111/j.1365-2796.2008.02024.x. PMID 19017170
- [Background] Carnio J, Miller PD Jr. Increasing the amount of attached gingiva using a modified apically repositioned flap. J Periodontol. 1999 Sep;70(9):1110-7. doi: 10.1902/jop.1999.70.9.1110. PMID 10505814
- [Background] Carnio J, Camargo PM, Passanezi E. Increasing the apico-coronal dimension of attached gingiva using the modified apically repositioned flap technique: a case series with a 6-month follow-up. J Periodontol. 2007 Sep;78(9):1825-30. doi: 10.1902/jop.2007.060414. PMID 17760555
- [Background] Buemi M, Galeano M, Sturiale A, Ientile R, Crisafulli C, Parisi A, Catania M, Calapai G, Impala P, Aloisi C, Squadrito F, Altavilla D, Bitto A, Tuccari G, Frisina N. Recombinant human erythropoietin stimulates angiogenesis and healing of ischemic skin wounds. Shock. 2004 Aug;22(2):169-73. doi: 10.1097/01.shk.0000133591.47776.bd. PMID 15257091